CLINICAL TRIAL: NCT07215611
Title: Financial Toxicity in Patients With Resected Soft Tissue and Bone Sarcomas
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-1156; NCI-2025-07460 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-10-09; First posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Bone Sarcomas; Financial Toxicity
MeSH Terms: conditions — Bone Neoplasms; Financial Stress | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: data collection — data collection from electronic health records

SUMMARY:
To learn about the financial stress patients undergoing surgery to treat orthopedic cancer experience because of the costs of cancer care, and to learn about the effects of financial stress on participants quality of life.

DETAILED DESCRIPTION:
Measure the prevalence of financial toxicity and the severity of it in orthopaedic oncology patients undergoing surgical intervention using an objective, validated instrument. Secondary objectives include identifying socioeconomic and demographic risk factors for financial toxicity and evaluating clinicopathologic characteristics that may worsen financial stress in this population.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are seen preoperatively at our institution before surgery for primary malignant bone tumor or primary malignant soft tissue tumor will be identified.
* Adult orthopedic oncology patients. Stratified by diagnosis of primary malignant bone tumor and primary malignant soft tissue tumor.

Exclusion Criteria

• Non-English subjects will not be recruited. Subjects are required to be able to read/write in English.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2028-10-02 (Estimated); Study Completion 2030-10-02 (Estimated)

PRIMARY OUTCOMES:
Questionnaires | Through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shalin S Patel, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org